CLINICAL TRIAL: NCT05207150
Title: Continuous Rhythm Monitoring With Implantable Cardiac Monitors And Wearable Devices With Real-time Smartphone Alerts During AF Episodes
Acronym: SMART-ALERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Tim Betts MD MBChB FRCP, Primary Investigator, Oxford University Hospitals NHS Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15634
Record Dates: First submitted 2021-12-12; First posted 2022-01-26 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation
Keywords: AF; Apple Watch; CART-I ring; LINQ II; Wearable
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LINQ II/Apple Watch Series 6 (Active Comparator)
  Interventions: Device: LINQII/Apple Watch Series 6
- LINQII/SkyLabs CART-I ring (Active Comparator)
  Interventions: Device: LINQII/SkyLabs CART-I ring

INTERVENTIONS:
Device: LINQII/Apple Watch Series 6 — LINQ II will be implanted and in the first 3 months it will send alerts to participants' smartphones if it detects an AF episode longer than 30 minutes. After 3 months, participants will wear an Apple Watch Series 6 for another 3 months. The LINQ II ICM will continue to detect and record AF episodes and will be used to validate the AF detection accuracy by the wearable devices but it will no longer send alerts during AF episodes. Instead, the wearable device (Apple Watch) will send a real-time alert to participants during AF episodes longer than 30 minutes and participants will use the appropriate smartphone app to acknowledge they have received the alert.
  Arms: LINQ II/Apple Watch Series 6
Device: LINQII/SkyLabs CART-I ring — LINQ II will be implanted and in the first 3 months it will send alerts to participants' smartphones if it detects an AF episode longer than 30 minutes. After 3 months, participants will wear a SkyLabs CART-I ring for another 3 months. The LINQ II ICM will continue to detect and record AF episodes and will be used to validate the AF detection accuracy by the wearable devices but it will no longer send alerts during AF episodes. Instead, the wearable device (CART-I ring) will send a real-time alert to participants during AF episodes longer than 30 minutes and participants will use the appropriate smartphone app to acknowledge they have received the alert.
  Arms: LINQII/SkyLabs CART-I ring

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia affecting 1.3 million people in the UK. AF causes an irregular and fast heartbeat, which makes the heart pump poorly. As a result, blood clots may form inside the heart and, if they travel to the brain, can lead to an AF-related stroke. Patients with AF have a risk of stroke five-times higher than patients with normal rhythm.

Anticoagulants make the blood less likely to clot and, thus, reduce the chances of an AF-related stroke. For most people, once anticoagulation is started it must be taken for the rest of their lives irrespective of the amount of AF someone has. However, anticoagulants make patients more prone to bleeding.

New studies have reported a lower stroke risk in patients with short and infrequent AF episodes. If there are long time gaps in between AF episodes, short periods of anticoagulation around the time of AF may be enough to avoid clots from forming and reducing the overall risk of bleeding. To use anticoagulants only when needed will require an accurate and reliable way to detect AF when it occurs and alert patients. New technologies, such as small heart monitors placed under the skin, watches and rings, can track the heart rhythm continuously and send real-time alerts to patients via mobile phone message if AF is detected.

The purpose of this study is to investigate if implantable cardiac monitors (LINQ II) and wearable devices (Apple Watch and CART-I ring) can detect AF episodes, send real-time alerts to patients and who will respond to these alerts within a short timeframe. The investigators will recruit 50 patients and follow them for six months. All participants will receive a LINQ II and a wearable device.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Male or Female aged 18 years or above.
* Paroxysmal AF with symptoms, Holter recording and/or implantable device evidence of >1 but <15 episodes of AF in the last 3 months.
* Persistent AF scheduled for repeat cardioversion (i.e. having had at least one prior cardioversion).
* Currently have an Apple IOS or Android smartphone.

Exclusion Criteria:

* Diagnosis of permanent AF.
* Contra-indications for implantable cardiac monitor.
* Visual or physical impairment that prevents ability to read and acknowledge smartphone/watch notifications.
* Unable to comply with the follow-up schedule.
* Do not have Apple IOS or android smartphone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
To assess the performance of the LINQ II™ ICM in sending real-time alerts to participants' smartphone and to Carelink (physicians web portal) during AF episodes longer than 30 minutes | During follow-up (6 months)
  Percentage of successful alerts sent by the LINQII™ ICM.

SECONDARY OUTCOMES:
To study the diagnostic accuracy of the Apple Watch and the Skylabs CART-I ring in the detection of AF episodes . | During the follow-up period (6 month)Apple Watch and Skylabs CART-I ring sensitivity, specificity, positive and negative predictive for AF episodes longer than 30 minutes.
  Apple Watch and Skylabs CART-I ring diagnostic accuracy for AF episodes longer than 30 minutes compared to the LINQ II™ ICM (gold standard).
To assess the performance of the Apple Watch and the Skylabs CART-I ring in sending real-time alerts to their smartphone apps and participants' engagement. | During follow-up (6 months)
  Percentage of successful alerts sent by the Apple Watch and Skylabs CART-I ring.
To study participants' compliance wih the Apple Watch and the Skylabs CART-I ring | During follow-up (6 months)
  Percentage of time the wearable devices have been used and comparison between different modalities will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Betts, MD MBChB FRCP, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Oxford Univeristy Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided